CLINICAL TRIAL: NCT03654885
Title: XEN-45 Gel Stent Versus Trabeculectomy in Glaucoma: Gold-Standard Pathway Study (GPS)
Acronym: XEN GPS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CMO-US-EYE-0600
Record Dates: First submitted 2018-08-23; First posted 2018-08-31 (Actual); Results first posted 2022-07-21 (Actual); Last update posted 2022-07-21 (Actual); Status verified 2022-06

CONDITIONS: Glaucoma
MeSH Terms: conditions — Glaucoma | interventions — Trabeculectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- XEN-45 Gel Stent (Active Comparator): Participants underwent at least one preoperative visit and had XEN-45 gel stent implantation on Day 0 (The day of surgery).
  Interventions: Device: XEN-45 Gel Stent
- Trabeculectomy (Active Comparator): Participants underwent at least one preoperative visit and had trabeculectomy as per standard of care in each investigative center on Day 0 (The day of surgery).
  Interventions: Procedure: Trabeculectomy

INTERVENTIONS:
Device: XEN-45 Gel Stent — XEN-45 gel stent device implant
  Arms: XEN-45 Gel Stent
Procedure: Trabeculectomy — Trabeculectomy surgery
  Arms: Trabeculectomy

SUMMARY:
The purpose of this study is to compare the safety and efficacy of XEN-45 to trabeculectomy in participants with open angle glaucoma refractory to topical medical therapy.

DETAILED DESCRIPTION:
This is a multi-center, randomized, parallel group, prospective, open-label clinical trial to evaluate the ability of XEN-45 to reduce intraocular pressure (IOP) and reduce the amount of topical IOP-lowering medications in participants poorly controlled on topical therapy. The planned study duration is 12 months. Participants were to be screened for enrollment and eligible candidates were to be approached to ascertain interest in study participation. Eligible participants were to be randomized 2:1; resulting in approximately 95 eyes implanted with XEN-45 and 44 eyes received trabeculetomy by study end.

ELIGIBILITY:
Inclusion Criteria:

* Open-angle glaucoma where the intraocular pressure (IOP) is not controlled when using topical IOP-lowering glaucoma medication
* Best-corrected baseline Snellen visual acuity of 20/100 or better
* Visual field mean deviation no worse than -18.0 decibels (dB)
* Medicated IOP ≥15 millimeter of mercury (mm Hg) and ≤44 mm Hg
* Participants not anticipated to require any ocular surgery (e.g., cataract surgery) in either eye up to 3 months from the time of inclusion
* Area of healthy, free, and mobile conjunctiva in the target area (superior bulbar conjunctiva)
* Trabecular meshwork must be visible (with Shaffer angle grade ≥2 in the target quadrant)
* Failed ab-interno canal or suprachoroidal micro invasive glaucoma surgery (MIGS) procedures (such as i-Stent, gonioscopy-assisted transluminal trabeculotomy [GATT], Ab-interno canaloplasty [ABiC], Kahook dual blade goniotomy, etc.) are allowed ≥3 months before enrollment. CyPass® Micro-Stents were not allowed.

Exclusion Criteria:

* Participant has active neovascular, uveitic or angle recession glaucoma or any glaucoma associated with vascular disorders
* Participant has had prior ab externo incisional glaucoma surgery (such as trabeculectomy, viscocanalostomy, canaloplasty, tube shunts of any type, collagen implants, etc.), conjunctival filtering surgery, transscleral cycloablative procedures (such as cyclophotocoagulation, micro pulse cyclophotocoagulation, cryotherapy, ultrasound circular cyclocoagulation [UC3], etc.) or prior major conjunctival surgery (i.e., scleral buckle)
* Clinically significant inflammation or infection within 30 days before the preoperative visit (e.g., blepharitis, conjunctivitis, severe ocular surface disease, keratitis, uveitis, herpes simplex infection)
* Presence of conjunctival scarring or prior conjunctival surgery or other conjunctival pathologies (e.g., pterygium) in the target area
* History of corneal surgery, corneal opacities, or corneal disease
* Central corneal thickness ≤490 micrometer (μm) or ≥620μm
* Vitreous present in the anterior chamber
* Aphakic
* Participant has had prior intraocular surgery in either eye within ≤3 months before the preoperative visit (including phacoemulsification)
* History of complicated cataract surgery (e.g. with visual impairment, e.g. vitreous loss, anterior chamber intraocular lens [ACIOL], perhaps sutured intraocular lens [IOL] or scleral fixated IOL, prior cystoid macular edema [CME], etc.)
* Presence of intraocular silicone oil
* Active diabetic retinopathy, proliferative retinopathy, choroidal neovascularization, branch retinal vein occlusion, central retinal vein occlusion, geographic atrophy, or other ophthalmic disease or disorder that could confound study results or impaired episcleral venous drainage (e.g., Sturge-Weber or nanophthalmos, Axenfeld-Reiger, iridocorneal endothelial syndrome [ICE], etc.)
* Known or suspected allergy or sensitivity to drugs required for the protocol (including anesthesia), or any of the device components (e.g., bovine or porcine products, or glutaraldehyde)
* Pregnant or nursing women and those planning a pregnancy during the study period.
* Participation in another drug or device clinical trial concluding within 30 days before the preoperative visit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2021-05-13 (Actual); Study Completion 2021-05-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: ALLERGAN INC., Study Director — Allergan
Locations (35):
- United States (35):
  - Vold Vision /ID# 233677, Fayetteville, Arkansas
  - Retina Institute of California /ID# 233692, Arcadia, California
  - Angeles Eye Institute /ID# 233632, Culver City, California
  - Cha Medical Group Pc /Id# 233649, Los Angeles, California
  - Grutzmacher Lewis and Sierra Inc. /ID# 233654, Sacramento, California
  - University of Colorado Denver /ID# 233676, Denver, Colorado
  - Howard University Hospital /ID# 233615, Washington D.C., District of Columbia
  - Eye Surgery Associates /ID# 233638, Hollywood, Florida
  - Specialty Retina Center /ID# 233628, Weston, Florida
  - Georgia Eye Partners /ID# 233655, Atlanta, Georgia
  - Coastal Research Associates /ID# 233575, Roswell, Georgia
  - Tyrie Lee Jenkins MD Inc. /ID# 233674, Honolulu, Hawaii
  - Illinois Eye Center /ID# 233631, Peoria, Illinois
  - Stiles Eyecare Excellence /ID# 233583, Overland Park, Kansas
  - Advanced Glaucoma Specialists /ID# 233690, Reading, Massachusetts
  - Kellogg Eye Center University of Michigan health system /ID# 233651, Ann Arbor, Michigan
  - Mayo Clinic Jacksonville /ID# 233634, Saint Paul, Minnesota
  - Washington University in St. Louis /ID# 233599, St Louis, Missouri
  - Glaucoma associates/consultants of the capital region /ID# 233695, Slingerlands, New York
  - Carolina Eye Associates /ID# 233656, Southern Pines, North Carolina
  - Eye Care Associates Inc /ID# 233636, Youngstown, Ohio
  - Dean McGee Eye Institute /ID# 233595, Oklahoma City, Oklahoma
  - Ludwick Eye Center /ID# 233691, Chambersburg, Pennsylvania
  - Kremer Eye Center /Id# 233642, King of Prussia, Pennsylvania
  - Wills Eye Institute /ID# 233645, Philadelphia, Pennsylvania
  - university of Pittsburgh /ID# 233622, Pittsburgh, Pennsylvania
  - Carolinas Centers for Sight,PC /ID# 233606, Florence, South Carolina
  - Nashville Vision Associates /ID# 233644, Nashville, Tennessee
  - Glaucoma Associates of Texas /ID# 233587, Dallas, Texas
  - El Paso Eye Surgeons, P.A. /ID# 233584, El Paso, Texas
  - Houston Eye Associates /ID# 233621, Houston, Texas
  - Baylor College of Medicine - Baylor Medical Center /ID# 233612, Houston, Texas
  - Vistar Eye Center /ID# 233652, Roanoke, Virginia
  - SSM Health Dean Medical Group /ID# 233624, Madison, Wisconsin
  - The Eye Centers of Racine and Kenosha LTD /ID# 233657, Racine, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols and clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing, please refer to the link below.
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous, independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Use Agreement (DUA). For more information on the process, or to submit a request, visit the following link.
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- [Derived] Sheybani A, Vera V, Grover DS, Vold SD, Cotter F, Bedrood S, Sawhney G, Piette SD, Simonyi S, Gu X, Balaram M, Gallardo MJ. Gel Stent Versus Trabeculectomy: The Randomized, Multicenter, Gold-Standard Pathway Study (GPS) of Effectiveness and Safety at 12 Months. Am J Ophthalmol. 2023 Aug;252:306-325. doi: 10.1016/j.ajo.2023.03.026. Epub 2023 Mar 25. PMID 36972738
- See also: Related Info — http://rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One eye, the worse eye, from each participant was selected as the study eye. The worse eye was defined using the visual field mean deviation (MD) at baseline, with the worse eye having the most negative MD. In the case where the MD was the same in both eyes, to two decimal places, the worse eye is defined as the eye with the higher IOP.
Units Other Than Participants: eyes
Period: Overall Study
Arm/Group | XEN-45 Gel Stent | Trabeculectomy
Started | 107; 107 eyes (One eye, the worse eye, from each participant was selected as the study eye.) | 51; 51 eyes (One eye, the worse eye, from each participant was selected as the study eye.)
Intent-to-Treat (ITT) Population (Intent-to-Treat (ITT) Population included all enrolled eyes/participants that were randomized to and received study glaucoma surgery (XEN-45 or trabeculectomy). Analyses were based on the randomized surgery.) | 95; 95 eyes | 44; 44 eyes
Safety Population (Safety Population included all enrolled participants that have undergone study glaucoma surgery.) | 95; 95 eyes | 44; 44 eyes
Completed | 77; 77 eyes | 38; 38 eyes
Not Completed | 30; 30 eyes | 13; 13 eyes
Not completed — Randomized, Not Treated: Consent Withdrawn | 5 | 3
Not completed — Randomized, Not Treated: Investigators Decision (Unrelated to Adverse Event [AE]) | 0 | 3
Not completed — Randomized, Not Treated: Study on-hold due to Device Recall | 7 | 1
Not completed — Additional Glaucoma Surgery (Secondary Surgical Intervention [SSI]) | 7 | 1
Not completed — Additional Ophthalmic Surgery (Not for Intraocular pressure [IOP] Control) | 1 | 0
Not completed — Adverse Event in Study Eye | 3 | 0
Not completed — Consent Withdrawn | 1 | 0
Not completed — Death | 3 | 1
Not completed — Did Not Meet Inclusion Criteria (IC) Diagnosis of Ocular Hypertension (Dx OHT) | 0 | 1
Not completed — Lost to Follow-up | 3 | 3

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) Population included all enrolled eyes/participants that were randomized to and received study glaucoma surgery (XEN-45 or trabeculectomy). Analyses were based on the randomized surgery.
Groups:
- Total: Total of all reporting groups
Arm/Group | XEN-45 Gel Stent | Trabeculectomy | Total
Number analyzed (Participants) | 95 | 44 | 139
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.5 (9.64) | 69.4 (9.72) | 69.5 (9.63)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 19 | 60
  Male | 54 | 25 | 79
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 18 | 10 | 28
  Asian | 2 | 0 | 2
  Black or African American | 14 | 8 | 22
  White or Caucasian | 61 | 26 | 87
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Ethnicity data was not collected
Study Eye Intraocular Pressure (IOP) [Mean (Standard Deviation); unit: millimetre of mercury (mm Hg)] — IOP is a measurement of the fluid pressure inside the eye. The worse eye was selected as the study eye if both eyes meet the inclusion criteria. The worse eye was defined using the visual field MD at baseline, with the worse eye having the most negative MD. In the case where the MD was the same in both eyes, to two decimal places, the worse eye is defined as the eye with the higher IOP.
  millimetre of mercury (mm Hg) | 23.13 (5.817) | 22.56 (5.653) | 22.95 (5.751)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving at Least 20% Intraocular Pressure (IOP) Reduction (Improvement) From Baseline at Month 12 With Prespecified Caveats
Description: IOP is a measure of the fluid pressure inside the eye. In addition to achieving a 20% reduction of IOP from Baseline, the participants had to meet all of the following prespecified caveats at Month 12: no increase in the number of topical IOP-lowering medications compared to Baseline, no clinical hypotony, no loss of vision to count fingers or worse, and no secondary glaucoma surgical intervention.
Time Frame: Baseline (Preoperative) to Month 12
Population: ITT Population included all enrolled eyes/participants that were randomized to and received study glaucoma surgery (XEN-45 or trabeculectomy). Analyses were based on the randomized surgery.
Measure: Number; unit: percentage of participants
Arm/Group | XEN-45 Gel Stent | Trabeculectomy
Number analyzed (Participants) | 95 | 44
percentage of participants | 62.1 | 68.2
Statistical Analysis 1: Comparison: XEN-45 Gel Stent; Test type: Non-Inferiority — By assuming the margin of non-inferiority at 24%, the null hypothesis for this non-inferiority testing was to be set up as XEN implanted group (P1)-Trabeculectomy group (P2) ≤-0.24 versus the alternative hypothesis as P1-P2 >-0.24. Equivalently, non-inferiority of P1 to P2 was to be declared if the lower limit of the 2-sided confidence interval (CI) of the difference of the above endpoint between the two treatment groups computed using normal approximation was found to be greater than -24%; p = 0.487, Chi-squared; Percentage Difference = -6.1, 95% CI 2-sided [-22.9 to 10.8]

2. Secondary Outcome: Mean IOP Over Time
Description: IOP is a measurement of the fluid pressure inside the eye.
Time Frame: Baseline and Day 1, Weeks 1 and 2, Months 1, 3, 6, 9, and 12
Population: ITT Population included all enrolled eyes/participants that were randomized to and received study glaucoma surgery (XEN-45 or trabeculectomy). Analyses were based on the randomized surgery. Number analyzed is the number of participants with data available for analysis at the specified timepoints.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | XEN-45 Gel Stent | Trabeculectomy
Number analyzed (Participants) | 95 | 44
mm Hg
  Day 1: number analyzed (Participants) | 95 | 43
  Day 1 | 9.25 (4.710) | 15.00 (13.025)
  Week 1: number analyzed (Participants) | 90 | 43
  Week 1 | 11.27 (6.864) | 11.48 (7.323)
  Week 2: number analyzed (Participants) | 91 | 43
  Week 2 | 13.64 (8.363) | 11.53 (5.503)
  Month 1: number analyzed (Participants) | 94 | 43
  Month 1 | 13.72 (6.315) | 11.45 (5.645)
  Month 3: number analyzed (Participants) | 89 | 41
  Month 3 | 16.46 (7.407) | 11.59 (4.672)
  Month 6: number analyzed (Participants) | 81 | 41
  Month 6 | 14.86 (4.228) | 11.72 (5.242)
  Month 9: number analyzed (Participants) | 81 | 41
  Month 9 | 14.57 (4.221) | 11.02 (3.535)
  Month 12: number analyzed (Participants) | 78 | 38
  Month 12 | 14.43 (4.060) | 11.83 (3.525)

3. Secondary Outcome: Change From Baseline in Mean IOP Over Time
Description: IOP is a measurement of the fluid pressure inside the eye.
Time Frame: Baseline and Day 1, Weeks 1 and 2, Months 1, 3, 6, 9, and 12
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | XEN-45 Gel Stent | Trabeculectomy
Number analyzed (Participants) | 95 | 44
mm Hg
  Change From Baseline at Day 1: number analyzed (Participants) | 95 | 43
  Change From Baseline at Day 1 | -13.63 (0.645) | -7.82 (0.958)
  Change From Baseline at Week 1: number analyzed (Participants) | 90 | 43
  Change From Baseline at Week 1 | -11.56 (0.660) | -11.34 (0.958)
  Change From Baseline at Week 2: number analyzed (Participants) | 91 | 43
  Change From Baseline at Week 2 | -9.26 (0.657) | -11.29 (0.958)
  Change From Baseline at Month 1: number analyzed (Participants) | 94 | 43
  Change From Baseline at Month 1 | -9.15 (0.648) | -11.37 (0.958)
  Change From Baseline at Month 3: number analyzed (Participants) | 89 | 41
  Change From Baseline at Month 3 | -6.35 (0.663) | -11.09 (0.977)
  Change From Baseline at Month 6: number analyzed (Participants) | 81 | 41
  Change From Baseline at Month 6 | -7.94 (0.690) | -10.95 (0.978)
  Change From Baseline at Month 9: number analyzed (Participants) | 81 | 41
  Change From Baseline at Month 9 | -8.19 (0.690) | -11.72 (0.978)
  Change From Baseline at Month 12: number analyzed (Participants) | 78 | 38
  Change From Baseline at Month 12 | -8.25 (0.701) | -11.02 (1.009)
Statistical Analysis 1: Comparison: XEN-45 Gel Stent vs Trabeculectomy; Change From Baseline in Mean IOP Over Time: Day 1; Test type: Other — No formal hypothesis was planned. P-value for treatment differences was provided for reference; p < 0.001, Mixed Model for Repeated Measures — Mixed Model for Repeated Measures (MMRM) model with treatment and time as the factors, treatment by time interaction and Baseline as the covariate variables were used for analysis; Percentage Difference = -5.81, 95% CI 2-sided [-8.074 to -3.538], Standard Error of Mean 1.155
Statistical Analysis 2: Comparison: XEN-45 Gel Stent vs Trabeculectomy; Change From Baseline in Mean IOP Over Time: Week 1; Test type: Other — No formal hypothesis was planned. P-value for treatment differences was provided for reference; p = 0.851, Mixed Model for Repeated Measures — MMRM model with treatment and time as the factors, treatment by time interaction and Baseline as the covariate variables were used for analysis; Percentage Difference = -0.22, 95% CI 2-sided [-2.503 to 2.066], Standard Error of Mean 1.163
Statistical Analysis 3: Comparison: XEN-45 Gel Stent vs Trabeculectomy; Change From Baseline in Mean IOP Over Time: Week 2; Test type: Other — No formal hypothesis was planned. P-value for treatment differences was provided for reference; p = 0.081, Mixed Model for Repeated Measures — [p-value comment as in outcome 3, analysis 2]; Percentage Difference = 2.03, 95% CI 2-sided [-0.253 to 4.309], Standard Error of Mean 1.162
Statistical Analysis 4: Comparison: XEN-45 Gel Stent vs Trabeculectomy; Change From Baseline in Mean IOP Over Time: Month 1; Test type: Other — No formal hypothesis was planned. P-value for treatment differences was provided for reference; p = 0.056, Mixed Model for Repeated Measures — [p-value comment as in outcome 3, analysis 2]; Percentage Difference = 2.21, 95% CI 2-sided [-0.059 to 4.484], Standard Error of Mean 1.157
Statistical Analysis 5: Comparison: XEN-45 Gel Stent vs Trabeculectomy; Change From Baseline in Mean IOP Over Time: Month 3; Test type: Other — No formal hypothesis was planned. P-value for treatment differences was provided for reference; p < 0.001, Mixed Model for Repeated Measures — [p-value comment as in outcome 3, analysis 2]; Percentage Difference = 4.74, 95% CI 2-sided [2.416 to 7.054], Standard Error of Mean 1.181
Statistical Analysis 6: Comparison: XEN-45 Gel Stent vs Trabeculectomy; Change From Baseline in Mean IOP Over Time: Month 6; Test type: Other — No formal hypothesis was planned. P-value for treatment differences was provided for reference; p = 0.012, Mixed Model for Repeated Measures — [p-value comment as in outcome 3, analysis 2]; Percentage Difference = 3.01, 95% CI 2-sided [0.657 to 5.358], Standard Error of Mean 1.197
Statistical Analysis 7: Comparison: XEN-45 Gel Stent vs Trabeculectomy; Change From Baseline in Mean IOP Over Time: Month 9; Test type: Other — No formal hypothesis was planned. P-value for treatment differences was provided for reference; p = 0.003, Mixed Model for Repeated Measures — [p-value comment as in outcome 3, analysis 2]; Percentage Difference = 3.53, 95% CI 2-sided [1.182 to 5.883], Standard Error of Mean 1.197
Statistical Analysis 8: Comparison: XEN-45 Gel Stent vs Trabeculectomy; Change From Baseline in Mean IOP Over Time: Month 12; Test type: Other — No formal hypothesis was planned. P-value for treatment differences was provided for reference; p = 0.024, Mixed Model for Repeated Measures — [p-value comment as in outcome 3, analysis 2]; Percentage Difference = 2.77, 95% CI 2-sided [0.358 to 5.183], Standard Error of Mean 1.229

4. Secondary Outcome: Mean Number of Topical IOP-Lowering Medications Over Time
Description: IOP is a measurement of the fluid pressure inside the eye. Topical IOP-lowering medication classes included: prostaglandin analogues, beta adrenergic antagonists, carbonic anhydrase inhibitors,alpha adrenergic agonists, pilocarpine, and combinations of these treatments.
Time Frame: Baseline and Day 1, Weeks 1 and 2, Months 1, 3, 6, 9, and 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: medications
Arm/Group | XEN-45 Gel Stent | Trabeculectomy
Number analyzed (Participants) | 95 | 44
medications
  Day 1 | 0.2 (0.51) | 0.3 (0.53)
  Week 1: number analyzed (Participants) | 94 | 43
  Week 1 | 0.3 (0.77) | 0.3 (0.73)
  Week 2: number analyzed (Participants) | 94 | 43
  Week 2 | 0.3 (0.64) | 0.2 (0.53)
  Month 1: number analyzed (Participants) | 94 | 43
  Month 1 | 0.3 (0.75) | 0.1 (0.52)
  Month 3: number analyzed (Participants) | 91 | 42
  Month 3 | 0.5 (0.89) | 0.1 (0.26)
  Month 6: number analyzed (Participants) | 82 | 41
  Month 6 | 0.6 (0.96) | 0.2 (0.58)
  Month 9: number analyzed (Participants) | 81 | 41
  Month 9 | 0.6 (1.09) | 0.2 (0.49)
  Month 12: number analyzed (Participants) | 87 | 41
  Month 12 | 0.6 (0.95) | 0.3 (0.50)

5. Secondary Outcome: Change From Baseline in Mean Number of Topical IOP-Lowering Medications Over Time
Description: as for outcome 4
Time Frame: Baseline and Day 1, Weeks 1 and 2, Months 1, 3, 6, 9, and 12
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: medications
Arm/Group | XEN-45 Gel Stent | Trabeculectomy
Number analyzed (Participants) | 95 | 44
medications
  Change From Baseline at Day 1 | -2.1 (0.08) | -2.0 (0.11)
  Change From Baseline at Week 1: number analyzed (Participants) | 94 | 43
  Change From Baseline at Week 1 | -2.0 (0.08) | -2.0 (0.11)
  Change From Baseline at Week 2: number analyzed (Participants) | 94 | 43
  Change From Baseline at Week 2 | -2.0 (0.08) | -2.1 (0.11)
  Change From Baseline at Month 1: number analyzed (Participants) | 94 | 43
  Change From Baseline at Month 1 | -2.0 (0.08) | -2.1 (0.11)
  Change From Baseline at Month 3: number analyzed (Participants) | 91 | 42
  Change From Baseline at Month 3 | -1.8 (0.08) | -2.2 (0.11)
  Change From Baseline at Month 6: number analyzed (Participants) | 82 | 41
  Change From Baseline at Month 6 | -1.7 (0.08) | -2.0 (0.11)
  Change From Baseline at Month 9: number analyzed (Participants) | 81 | 41
  Change From Baseline at Month 9 | -1.7 (0.08) | -2.0 (0.11)
  Change From Baseline at Month 12: number analyzed (Participants) | 87 | 41
  Change From Baseline at Month 12 | -1.7 (0.08) | -2.0 (0.11)
Statistical Analysis 1: Comparison: XEN-45 Gel Stent; Change from Baseline in Mean Number of Topical IOP-Lowering Medications Over Time: Day 1; Test type: Other — No formal hypothesis was planned. P-value for treatment differences was provided for reference; p = 0.505, Mixed Model for Repeated Measures — [p-value comment as in outcome 3, analysis 2]; Percentage Difference = -0.1, 95% CI 2-sided [-0.36 to 0.18], Standard Error of Mean 0.14
Statistical Analysis 2: Comparison: XEN-45 Gel Stent vs Trabeculectomy; Change from Baseline in Mean Number of Topical IOP-Lowering Medications Over Time: Week 1; Test type: Other — No formal hypothesis was planned. P-value for treatment differences was provided for reference; p = 0.949, Mixed Model for Repeated Measures — [p-value comment as in outcome 3, analysis 2]; Percentage Difference = 0.0, 95% CI 2-sided [-0.28 to 0.26], Standard Error of Mean 0.14
Statistical Analysis 3: Comparison: XEN-45 Gel Stent vs Trabeculectomy; Change from Baseline in Mean Number of Topical IOP-Lowering Medications Over Time: Week 2; Test type: Other — No formal hypothesis was planned. P-value for treatment differences was provided for reference; p = 0.581, Mixed Model for Repeated Measures — [p-value comment as in outcome 3, analysis 2]; Percentage Difference = 0.1, 95% CI 2-sided [-0.19 to 0.34], Standard Error of Mean 0.14
Statistical Analysis 4: Comparison: XEN-45 Gel Stent vs Trabeculectomy; Change from Baseline in Mean Number of Topical IOP-Lowering Medications Over Time: Month 1; Test type: Other — No formal hypothesis was planned. P-value for treatment differences was provided for reference; p = 0.302, Mixed Model for Repeated Measures — [p-value comment as in outcome 3, analysis 2]; Percentage Difference = 0.1, 95% CI 2-sided [-0.13 to 0.41], Standard Error of Mean 0.14
Statistical Analysis 5: Comparison: XEN-45 Gel Stent vs Trabeculectomy; Change from Baseline in Mean Number of Topical IOP-Lowering Medications Over Time: Month 3; Test type: Other — No formal hypothesis was planned. P-value for treatment differences was provided for reference; p = 0.005, Mixed Model for Repeated Measures — [p-value comment as in outcome 3, analysis 2]; Percentage Difference = 0.4, 95% CI 2-sided [0.12 to 0.66], Standard Error of Mean 0.14
Statistical Analysis 6: Comparison: XEN-45 Gel Stent vs Trabeculectomy; Change from Baseline in Mean Number of Topical IOP-Lowering Medications Over Time: Month 6; Test type: Other — No formal hypothesis was planned. P-value for treatment differences was provided for reference; p = 0.026, Mixed Model for Repeated Measures — [p-value comment as in outcome 3, analysis 2]; Percentage Difference = 0.3, 95% CI 2-sided [0.04 to 0.59], Standard Error of Mean 0.14
Statistical Analysis 7: Comparison: XEN-45 Gel Stent vs Trabeculectomy; Change from Baseline in Mean Number of Topical IOP-Lowering Medications Over Time: Month 9; Test type: Other — No formal hypothesis was planned. P-value for treatment differences was provided for reference; p = 0.010, Mixed Model for Repeated Measures — [p-value comment as in outcome 3, analysis 2]; Percentage Difference = 0.4, 95% CI 2-sided [0.09 to 0.64], Standard Error of Mean 0.14
Statistical Analysis 8: Comparison: XEN-45 Gel Stent vs Trabeculectomy; Change from Baseline in Mean Number of Topical IOP-Lowering Medications Over Time: Month 12; Test type: Other — No formal hypothesis was planned. P-value for treatment differences was provided for reference; p = 0.052, Mixed Model for Repeated Measures — [p-value comment as in outcome 3, analysis 2]; Percentage Difference = 0.3, 95% CI 2-sided [0.00 to 0.54], Standard Error of Mean 0.14

6. Secondary Outcome: Change From Baseline in Mean IOP at Month 12
Description: IOP is a measurement of the fluid pressure inside the eye.
Time Frame: Baseline (Preoperative) and Month 12
Population: ITT Population included all enrolled eyes/participants that were randomized to and received study glaucoma surgery (XEN-45 or trabeculectomy). Analyses were based on the randomized surgery Overall number analyzed are the number of participants with data available for analyses.
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | XEN-45 Gel Stent | Trabeculectomy
Number analyzed (Participants) | 78 | 38
mm Hg | -8.25 (0.701) | -11.02 (1.009)
Statistical Analysis 1: Comparison: XEN-45 Gel Stent vs Trabeculectomy; Test type: Other — No formal hypothesis was planned. P-value for treatment differences was provided for reference; p = 0.024, Mixed Model for Repeated Measures — MMRM model with treatment and time as the factors, treatment by time interaction and baseline as the covariate variables was used for analysis; Least Square Mean Difference = 2.77, 95% CI 2-sided [0.358 to 5.183], Standard Error of Mean 1.229

7. Secondary Outcome: Change From Baseline in Mean Number of Topical IOP-Lowering Medications at Month 12
Description: IOP is a measurement of the fluid pressure inside the eye. Topical IOP-lowering medication classes included: prostaglandin analogues, beta adrenergic antagonists, carbonic anhydrase inhibitors, alpha adrenergic agonists, pilocarpine, and combinations of these treatments.
Time Frame: Baseline (Preoperative) and Month 12
Population: ITT Population included all enrolled eyes/participants that were randomized to and received study glaucoma surgery (XEN-45 or trabeculectomy). Analyses were based on the randomized surgery. Overall number analyzed are the number of participants with data available for analyses.
Measure: Least Squares Mean (Standard Error); unit: medications
Arm/Group | XEN-45 Gel Stent | Trabeculectomy
Number analyzed (Participants) | 87 | 41
medications | -1.7 (0.08) | -2.0 (0.11)
Statistical Analysis 1: Comparison: XEN-45 Gel Stent vs Trabeculectomy; Test type: Other — No formal hypothesis was planned. P-value for treatment differences was provided for reference; p = 0.052, Mixed Model for Repeated Measures — [p-value comment as in outcome 6, analysis 1]; Least Square Mean Difference = 0.3, 95% CI 2-sided [0.00 to 0.54], Standard Error of Mean 0.14

8. Secondary Outcome: Change in Mean IOP From Preoperative Baseline Over Time in Participants With Eyes With Baseline IOP ≤18 mm Hg
Description: IOP is a measurement of the fluid pressure inside the eye.
Time Frame: Baseline (Preoperative) and Month 12
Population: ITT Population included all enrolled eyes/participants that were randomized to and received study glaucoma surgery (XEN-45 or trabeculectomy). Analyses were based on the randomized surgery. Overall number analyzed are the number of participants with Baseline IOP ≤18 mmHg in the ITT population and data available for analyses.
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | XEN-45 Gel Stent | Trabeculectomy
Number analyzed (Participants) | 18 | 9
mm Hg | -2.83 (1.281) | -4.61 (1.801)
Statistical Analysis 1: Comparison: XEN-45 Gel Stent vs Trabeculectomy; Test type: Other — No formal hypothesis was planned. P-value for treatment differences was provided for reference; p = 0.421, Mixed model repeated measures — [p-value comment as in outcome 6, analysis 1]; Least Square Mean Difference = 1.79, 95% CI 2-sided [-2.579 to 6.151], Standard Error of Mean 2.214

9. Secondary Outcome: Change in Number of Topical IOP-Lowering Medications From Preoperative Baseline to Month 12 in Participants With Eyes With Baseline IOP ≤18 mm Hg
Description: Topical IOP-lowering medication classes included: prostaglandin analogues, beta adrenergic antagonists, carbonic anhydrase inhibitors, alpha adrenergic agonists, pilocarpine, and combinations of these treatments.
Time Frame: Baseline (Preoperative) and Month 12
Population: as for outcome 8
Measure: Least Squares Mean (Standard Error); unit: medications
Arm/Group | XEN-45 Gel Stent | Trabeculectomy
Number analyzed (Participants) | 20 | 11
medications | -1.8 (0.15) | -2.1 (0.20)
Statistical Analysis 1: Comparison: XEN-45 Gel Stent vs Trabeculectomy; Test type: Other — No formal hypothesis was planned. P-value for treatment differences was provided for reference; p = 0.180, Mixed Model for Repeated Measures — [p-value comment as in outcome 6, analysis 1]; Least Square Mean Difference = 0.3, 95% CI 2-sided [-0.16 to 0.84], Standard Error of Mean 0.25

10. Secondary Outcome: Percentage of Participants Achieving Specific IOP Targets at Month 12
Description: IOP is a measurement of the fluid pressure inside the eye. Specific IOP targets included following IOP values (in mm Hg): ≤18, ≤17, ≤16, ≤15, ≤14, ≤13, ≤12 mm Hg.
Time Frame: Month 12
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Units Other Than Participants: eyes
Arm/Group | XEN-45 Gel Stent | Trabeculectomy
Number analyzed (Participants) | 95 | 44
Number analyzed (eyes) | 95 | 44
percentage of participants
  IOP Value of ≤18 mm Hg | 68.4 | 84.1
  IOP Value of ≤17 mm Hg | 64.2 | 79.5
  IOP Value of ≤16 mm Hg | 62.1 | 79.5
  IOP Value of ≤15 mm Hg | 55.8 | 72.7
  IOP Value of ≤14 mm Hg | 50.5 | 63.6
  IOP Value of ≤13 mm Hg | 36.8 | 56.8
  IOP Value of ≤12 mm Hg | 30.5 | 43.2
Statistical Analysis 1: Comparison: XEN-45 Gel Stent vs Trabeculectomy; Percentage of Participants Achieving Specific IOP Targets at Month 12: IOP Value of ≤18 mmHg; Test type: Other — No formal hypothesis was planned. P-value for treatment differences was provided for reference; p = 0.064, Fisher Exact; Percentage Difference = -15.7, 95% CI 2-sided [-33.0 to 2.3]
Statistical Analysis 2: Comparison: XEN-45 Gel Stent vs Trabeculectomy; Percentage of Participants Achieving Specific IOP Targets at Month 12: IOP Value of ≤17 mmHg; Test type: Other — No formal hypothesis was planned. P-value for treatment differences was provided for reference; p = 0.078, Fisher Exact; Percentage Difference = -15.3, 95% CI 2-sided [-32.7 to 2.5]
Statistical Analysis 3: Comparison: XEN-45 Gel Stent vs Trabeculectomy; Percentage of Participants Achieving Specific IOP Targets at Month 12: IOP Value of ≤16 mmHg; Test type: Other — No formal hypothesis was planned. P-value for treatment differences was provided for reference; p = 0.051, Fisher Exact; Percentage Difference = -17.4, 95% CI 2-sided [-34.7 to 0.4]
Statistical Analysis 4: Comparison: XEN-45 Gel Stent vs Trabeculectomy; Percentage of Participants Achieving Specific IOP Targets at Month 12: IOP Value of ≤15 mmHg; Test type: Other — No formal hypothesis was planned. P-value for treatment differences was provided for reference; p = 0.064, Fisher Exact; Percentage Difference = -16.9, 95% CI 2-sided [-34.1 to 1.0]
Statistical Analysis 5: Comparison: XEN-45 Gel Stent vs Trabeculectomy; Percentage of Participants Achieving Specific IOP Targets at Month 12: IOP Value of ≤14 mm Hg; Test type: Other — No formal hypothesis was planned. P-value for treatment differences was provided for reference; p = 0.200, Fisher Exact; Percentage Difference = -13.1, 95% CI 2-sided [-30.5 to 4.8]
Statistical Analysis 6: Comparison: XEN-45 Gel Stent vs Trabeculectomy; Percentage of Participants Achieving Specific IOP Targets at Month 12: IOP Value of ≤13 mm Hg; Test type: Other — No formal hypothesis was planned. P-value for treatment differences was provided for reference; p = 0.042, Fisher Exact; Percentage Difference = -20.0, 95% CI 2-sided [-37.1 to -2.0]
Statistical Analysis 7: Comparison: XEN-45 Gel Stent vs Trabeculectomy; Percentage of Participants Achieving Specific IOP Targets at Month 12: IOP Value of ≤12 mm Hg; Test type: Other — No formal hypothesis was planned. P-value for treatment differences was provided for reference; p = 0.180, Fisher Exact; Percentage Difference = -12.7, 95% CI 2-sided [-30.1 to 5.2]

11. Secondary Outcome: Percentage of Participants Achieving Specific Percentage IOP Lower Targets From Baseline at Month 12
Description: IOP is a measurement of fluid pressure inside the eye. Specific percentage IOP lower targets included ≥25%, ≥30%, ≥35%, ≥40% ≥45%, and ≥50% IOP reduction.
Time Frame: Baseline (Preoperative) to Month 12
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Units Other Than Participants: eyes
Arm/Group | XEN-45 Gel Stent | Trabeculectomy
Number analyzed (Participants) | 95 | 44
Number analyzed (eyes) | 95 | 44
percentage of participants
  ≥25% IOP Reduction | 60.0 | 63.6
  ≥30% IOP Reduction | 48.4 | 61.4
  ≥35% IOP Reduction | 41.1 | 61.4
  ≥40% IOP Reduction | 35.8 | 54.5
  ≥45% IOP Reduction | 25.3 | 43.2
  ≥50% IOP Reduction | 22.1 | 43.2
Statistical Analysis 1: Comparison: XEN-45 Gel Stent vs Trabeculectomy; Percentage of Participants Achieving Specific Percentage IOP Lower Targets From Baseline at Month 12: ≥25% IOP Reduction; Test type: Other — No formal hypothesis was planned. P-value for treatment differences was provided for reference; p = 0.712, Fisher Exact; Percentage Difference = -3.6, 95% CI 2-sided [-21.3 to 14.2]
Statistical Analysis 2: Comparison: XEN-45 Gel Stent vs Trabeculectomy; Percentage of Participants Achieving Specific Percentage IOP Lower Targets From Baseline at Month 12: ≥30% IOP Reduction; Test type: Other — No formal hypothesis was planned. P-value for treatment differences was provided for reference; p = 0.201, Fisher Exact; Percentage Difference = -12.9, 95% CI 2-sided [-30.3 to 5.0]
Statistical Analysis 3: Comparison: XEN-45 Gel Stent vs Trabeculectomy; Percentage of Participants Achieving Specific Percentage IOP Lower Targets From Baseline at Month 12: ≥35% IOP Reduction; Test type: Other — No formal hypothesis was planned. P-value for treatment differences was provided for reference; p = 0.030, Fisher Exact; Percentage Difference = -20.3, 95% CI 2-sided [-37.3 to -2.3]
Statistical Analysis 4: Comparison: XEN-45 Gel Stent vs Trabeculectomy; Percentage of Participants Achieving Specific Percentage IOP Lower Targets From Baseline at Month 12: ≥40% IOP Reduction; Test type: Other — No formal hypothesis was planned. P-value for treatment differences was provided for reference; p = 0.043, Fisher Exact; Percentage Difference = -18.8, 95% CI 2-sided [-36.0 to -0.8]
Statistical Analysis 5: Comparison: XEN-45 Gel Stent vs Trabeculectomy; Percentage of Participants Achieving Specific Percentage IOP Lower Targets From Baseline at Month 12: ≥45% IOP Reduction; Test type: Other — No formal hypothesis was planned. P-value for treatment differences was provided for reference; p = 0.048, Fisher Exact; Percentage Difference = -17.9, 95% CI 2-sided [-35.1 to 0.0]
Statistical Analysis 6: Comparison: XEN-45 Gel Stent vs Trabeculectomy; Percentage of Participants Achieving Specific Percentage IOP Lower Targets From Baseline at Month 12: ≥50% IOP Reduction; Test type: Other — No formal hypothesis was planned. P-value for treatment differences was provided for reference; p = 0.015, Fisher Exact; Percentage Difference = -21.1, 95% CI 2-sided [-38.1 to -3.2]

12. Secondary Outcome: Percentage of Participants Achieving at Least a 20% IOP Reduction and Specific IOP Targets on Same or Lower Number of Topical IOP-Lowering Medications at Month 12
Description: IOP is a measurement of fluid pressure inside the eye. Specific IOP targets included following IOP values (in mm Hg): ≤18, ≤17, ≤16, ≤15, ≤14, ≤13, ≤12 mm Hg.
Time Frame: Baseline (Preoperative) and Month 12
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | XEN-45 Gel Stent | Trabeculectomy
Number analyzed (Participants) | 95 | 44
percentage of participants
  IOP Target ≤18 mm Hg | 61.1 | 72.7
  IOP Target ≤17 mm Hg | 58.9 | 70.5
  IOP Target ≤16 mm Hg | 56.8 | 70.5
  IOP Target ≤15 mm Hg | 55.8 | 70.5
  IOP Target ≤14 mm Hg | 50.5 | 61.4
  IOP Target ≤13 mm Hg | 36.8 | 54.5
  IOP Target ≤12 mm Hg | 30.5 | 43.2
Statistical Analysis 1: Comparison: XEN-45 Gel Stent vs Trabeculectomy; Percentage of Participants Achieving at Least a 20% IOP Reductions and Specific IOP Targets on Same or Lower Number of Topical IOP-Lowering Medications at Month 12- IOP Target ≤18 mm Hg; Test type: Other — No formal hypothesis was planned. P-value for treatment differences was provided for reference; p = 0.252, Fisher Exact; Percentage Difference = -11.7, 95% CI 2-sided [-29.0 to 6.3]
Statistical Analysis 2: Comparison: XEN-45 Gel Stent vs Trabeculectomy; Percentage of Participants Achieving at Least a 20% IOP Reductions and Specific IOP Targets on Same or Lower Number of Topical IOP-Lowering Medications at Month 12- IOP Target ≤17 mmHg; Test type: Other — No formal hypothesis was planned. P-value for treatment differences was provided for reference; p = 0.258, Fisher Exact; Percentage Difference = -11.5, 95% CI 2-sided [-28.9 to 6.5]
Statistical Analysis 3: Comparison: XEN-45 Gel Stent vs Trabeculectomy; Percentage of Participants Achieving at Least a 20% IOP Reductions and Specific IOP Targets on Same or Lower Number of Topical IOP-Lowering Medications at Month 12- IOP Target ≤16 mm Hg; Test type: Other — No formal hypothesis was planned. P-value for treatment differences was provided for reference; p = 0.139, Fisher Exact; Percentage Difference = -13.6, 95% CI 2-sided [-30.9 to 4.4]
Statistical Analysis 4: Comparison: XEN-45 Gel Stent vs Trabeculectomy; Percentage of Participants Achieving at Least a 20% IOP Reductions and Specific IOP Targets on Same or Lower Number of Topical IOP-Lowering Medications at Month 12- IOP Target ≤15 mm Hg; Test type: Other — No formal hypothesis was planned. P-value for treatment differences was provided for reference; p = 0.136, Fisher Exact; Percentage Difference = -14.7, 95% CI 2-sided [-32.0 to 3.3]
Statistical Analysis 5: Comparison: XEN-45 Gel Stent vs Trabeculectomy; Percentage of Participants Achieving at Least a 20% IOP Reductions and Specific IOP Targets on Same or Lower Number of Topical IOP-Lowering Medications at Month 12- IOP Target ≤14 mm Hg; Test type: Other — No formal hypothesis was planned. P-value for treatment differences was provided for reference.%; p = 0.274, Fisher Exact; Percentage Difference = -10.8, 95% CI 2-sided [-28.2 to 7.1]
Statistical Analysis 6: Comparison: XEN-45 Gel Stent vs Trabeculectomy; Percentage of Participants Achieving at Least a 20% IOP Reductions and Specific IOP Targets on Same or Lower Number of Topical IOP-Lowering Medications at Month 12- IOP Target ≤13 mm Hg; Test type: Other — No formal hypothesis was planned. P-value for treatment differences was provided for reference; p = 0.065, Fisher Exact; Percentage Difference = -17.7, 95% CI 2-sided [-35.0 to 0.3]
Statistical Analysis 7: Comparison: XEN-45 Gel Stent vs Trabeculectomy; Percentage of Participants Achieving at Least a 20% IOP Reductions and Specific IOP Targets on Same or Lower Number of Topical IOP-Lowering Medications at Month 12- IOP Target ≤12 mmHg; Test type: Other — No formal hypothesis was planned. P-value for treatment differences was provided for reference; p = 0.180, Fisher Exact; Percentage Difference = -12.7, 95% CI 2-sided [-30.1 to 5.2]

13. Secondary Outcome: Percentage of Participants With Needlings Performed
Description: Needling of eye involves breaking down the wall of the scar using a fine needle to improve the drainage of fluid inside the eye.
Time Frame: Up to Month 12
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | XEN-45 Gel Stent | Trabeculectomy
Number analyzed (Participants) | 95 | 44
percentage of participants | 23.2 | 18.2

14. Secondary Outcome: Mean Number of Needlings Per Eye
Description: as for outcome 13
Time Frame: Up to Month 12
Population: ITT Population included all enrolled eyes/participants that were randomized to and received study glaucoma surgery (XEN-45 or trabeculectomy). Analyses were based on the randomized surgery. Overall number analyzed are the number of participants who had needlings with evaluable assessment at a specific timepoint.
Measure: Mean (Standard Deviation); unit: needlings
Arm/Group | XEN-45 Gel Stent | Trabeculectomy
Number analyzed (Participants) | 22 | 8
needlings | 1.7 (1.03) | 1.4 (0.74)

15. Secondary Outcome: Percentage of Eyes Achieving at Least a 20% Reduction in IOP at Month 12 on the Same or Fewer Topical IOP-lowering Medications in Participants Who Had Needlings
Description: IOP is a measurement of fluid pressure inside the eye. Topical IOP-lowering medication classes include: prostaglandin analogues, beta adrenergic antagonists, carbonic anhydrase inhibitors, alpha adrenergic agonists, pilocarpine, and combinations of these treatments.
Time Frame: Month 12
Population: ITT Population included all enrolled eyes/participants that were randomized to and received study glaucoma surgery (XEN-45 or trabeculectomy). Analyses were based on the randomized surgery. Overall number analyzed are the number of participants who had needlings with evaluable assessment.
Measure: Number; unit: percentage of eyes
Units Other Than Participants: Eyes
Arm/Group | XEN-45 Gel Stent | Trabeculectomy
Number analyzed (Participants) | 16 | 7
Number analyzed (Eyes) | 16 | 7
percentage of eyes | 87.5 | 85.7
Statistical Analysis 1: Comparison: XEN-45 Gel Stent vs Trabeculectomy; Test type: Other — No formal hypothesis was planned. P-value for treatment differences was provided for reference; p = 1.000, Fisher Exact; Percentage Difference = 1.8, 95% CI 2-sided [-41.6 to 44.1]

16. Secondary Outcome: Percentage of Eyes Not Using Any Topical IOP-lowering Medications in Participants Who Had Needlings
Description: as for outcome 9
Time Frame: Month 12
Population: as for outcome 15
Measure: Number; unit: percentage of eyes
Units Other Than Participants: Eyes
Arm/Group | XEN-45 Gel Stent | Trabeculectomy
Number analyzed (Participants) | 21 | 8
Number analyzed (Eyes) | 21 | 8
percentage of eyes | 42.9 | 75.0
Statistical Analysis 1: Comparison: XEN-45 Gel Stent vs Trabeculectomy; Test type: Other — No formal hypothesis was planned. P-value for treatment differences was provided for reference; p = 0.215, Fisher Exact; Percentage Difference = -32.1, 95% CI 2-sided [-66.8 to 10.0]

17. Secondary Outcome: Percentage of Participants With Antifibrotic Use During Needling
Description: Antifibrotic use included mitomycin-C (MMC) which was standardized for both groups and administered according to physician training and practice.
Time Frame: Up to Month 12
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | XEN-45 Gel Stent | Trabeculectomy
Number analyzed (Participants) | 95 | 44
percentage of participants | 16.8 | 15.9

18. Secondary Outcome: Percentage of Participants Achieving Complete Success at Month 12
Description: Complete success was defined as IOP ≤18mm Hg, with 20% or greater IOP lowering from medicated Baseline, on no topical medications, and no clinical hypotony. The topical medication included any topical ophthalmic medication used on the study eye regardless of the indication and dosage.
Time Frame: Month 12
Population: ITT Population included all enrolled eyes/participants that were randomized to and received study glaucoma surgery (XEN-45 or trabeculectomy). Analyses were based on the randomized surgery. This outcome measure was analyzed among the participants without topical medication at Baseline Qualifying Visit. Number analyzed is the number of participants with data available for analysis at specific timepoint.
Measure: Number; unit: percentage of participants
Arm/Group | XEN-45 Gel Stent | Trabeculectomy
Number analyzed (Participants) | 95 | 44
percentage of participants | 44.2 | 59.1
Statistical Analysis 1: Comparison: XEN-45 Gel Stent vs Trabeculectomy; Test type: Other — No formal hypothesis was planned. P-value for treatment differences was provided for reference; p = 0.144, Fisher Exact; Percentage Difference = -14.9, 95% CI 2-sided [-32.2 to 3.1]

19. Secondary Outcome: Percentage of Participants Achieving Qualified Success at Month 12
Description: Qualified success was defined as IOP ≤18 mm Hg, with 20% or greater IOP lowering from medicated Baseline, taking topical medications at Baseline Qualifying Visit, no clinical hypotony. The topical medication included any topical ophthalmic medication used on the study eye regardless of the indication and dosage.
Time Frame: Month12
Population: ITT Population included all enrolled eyes/participants that were randomized to and received study glaucoma surgery (XEN-45 or trabeculectomy). Analyses were based on the randomized surgery. This outcome measure was analyzed among the participants with topical medication at Baseline Qualifying Visit. Number analyzed is the number of participants with data available for analysis at specific timepoint.
Measure: Number; unit: percentage of participants
Arm/Group | XEN-45 Gel Stent | Trabeculectomy
Number analyzed (Participants) | 95 | 44
percentage of participants | 62.1 | 72.7
Statistical Analysis 1: Comparison: XEN-45 Gel Stent vs Trabeculectomy; Test type: Other — No formal hypothesis was planned. P-value for treatment differences was provided for reference; p = 0.254, Fisher Exact; Percentage Difference = -10.6, 95% CI 2-sided [-28.0 to 7.3]

20. Secondary Outcome: Percentage of Participants Achieving Specific IOP Targets at Month 12 in Medication-free Eye
Description: IOP is a measurement of the fluid pressure inside the eye. Specific IOP targets included following IOP values (in mm Hg): ≤18, ≤17, ≤16, ≤15, ≤14, ≤13, ≤12 mm Hg. Medication-free eye at Month 12 was defined as no IOP-lowering medication was used to the study eye at Month 12.
Time Frame: Month 12
Population: ITT Population included all enrolled eyes/participants that were randomized to and received study glaucoma surgery (XEN-45 or trabeculectomy). Analyses were based on the randomized surgery. Overall number analyzed are the number of participants who were medication free at Month 12 with evaluable assessment.
Measure: Number; unit: percentage of participants
Arm/Group | XEN-45 Gel Stent | Trabeculectomy
Number analyzed (Participants) | 59 | 31
percentage of participants
  IOP Target ≤18 mm Hg | 79.7 | 87.1
  IOP Target ≤17 mm Hg | 74.6 | 87.1
  IOP Target ≤16 mm Hg | 71.2 | 87.1
  IOP Target ≤15 mm Hg | 64.4 | 83.9
  IOP Target ≤14 mm Hg | 59.3 | 80.6
  IOP Target ≤13 mm Hg | 47.5 | 71.0
  IOP Target ≤12 mm Hg | 37.3 | 58.1
Statistical Analysis 1: Comparison: XEN-45 Gel Stent vs Trabeculectomy; Percentage of Participants Achieving Specific IOP Targets at Month 12 in Medication-free Eye- IOP Target ≤18 mm Hg; Test type: Other — No formal hypothesis was planned. P-value for treatment differences was provided for reference; p = 0.563, Fisher Exact; Percentage Difference = -7.4, 95% CI 2-sided [-28.6 to 14.2]
Statistical Analysis 2: Comparison: XEN-45 Gel Stent vs Trabeculectomy; Percentage of Participants Achieving Specific IOP Targets at Month 12 in Medication-free Eye- IOP Target ≤17 mm Hg; Test type: Other — No formal hypothesis was planned. P-value for treatment differences was provided for reference; p = 0.188, Fisher Exact; Percentage Difference = -12.5, 95% CI 2-sided [-33.5 to 9.1]
Statistical Analysis 3: Comparison: XEN-45 Gel Stent vs Trabeculectomy; Percentage of Participants Achieving Specific IOP Targets at Month 12 in Medication-free Eye- IOP Target ≤16 mmHg; Test type: Other — No formal hypothesis was planned. P-value for treatment differences was provided for reference; p = 0.118, Fisher Exact; Percentage Difference = -15.9, 95% CI 2-sided [-36.7 to 5.6]
Statistical Analysis 4: Comparison: XEN-45 Gel Stent vs Trabeculectomy; Percentage of Participants Achieving Specific IOP Targets at Month 12 in Medication-free Eye- IOP Target ≤15 mm Hg; Test type: Other — No formal hypothesis was planned. P-value for treatment differences was provided for reference; p = 0.085, Fisher Exact; Percentage Difference = -19.5, 95% CI 2-sided [-40.2 to 2.1]
Statistical Analysis 5: Comparison: XEN-45 Gel Stent vs Trabeculectomy; Percentage of Participants Achieving Specific IOP Targets at Month 12 in Medication-free Eye- IOP Target ≤14 mm Hg; Test type: Other — No formal hypothesis was planned. P-value for treatment differences was provided for reference; p = 0.059, Fisher Exact; Percentage Difference = -21.3, 95% CI 2-sided [-42.0 to 0.4]
Statistical Analysis 6: Comparison: XEN-45 Gel Stent vs Trabeculectomy; Percentage of Participants Achieving Specific IOP Targets at Month 12 in Medication-free Eye- IOP Target ≤13 mm Hg; Test type: Other — No formal hypothesis was planned. P-value for treatment differences was provided for reference; p = 0.045, Fisher Exact; Percentage Difference = -23.5, 95% CI 2-sided [-43.9 to -1.4]
Statistical Analysis 7: Comparison: XEN-45 Gel Stent vs Trabeculectomy; Percentage of Participants Achieving Specific IOP Targets at Month 12 in Medication-free Eye- IOP Target ≤12 mm Hg; Test type: Other — No formal hypothesis was planned. P-value for treatment differences was provided for reference; p = 0.076, Fisher Exact; Percentage Difference = -20.8, 95% CI 2-sided [-41.3 to 1.1]

21. Secondary Outcome: Percentage of Participants Achieving Specific Percentage IOP Lower Targets From Baseline at Month 12 With Medication-free Eyes
Description: IOP is a measurement of the fluid pressure inside the eye. Specific percentage IOP lower targets included ≥25%, ≥30%, ≥35%, ≥40% ≥45%, and ≥50% IOP reduction. Medication-free eye at Month 12 was defined as no IOP-lowering medication was used to the study eye at Month 12.
Time Frame: Month 12
Population: as for outcome 7
Measure: Number; unit: percentage of participants
Arm/Group | XEN-45 Gel Stent | Trabeculectomy
Number analyzed (Participants) | 59 | 31
percentage of participants
  ≥25% IOP Reduction | 67.8 | 77.4
  ≥30% IOP Reduction | 57.6 | 77.4
  ≥35% IOP Reduction | 50.8 | 77.4
  ≥40% IOP Reduction | 44.1 | 67.7
  ≥45% IOP Reduction | 30.5 | 58.1
  ≥50% IOP Reduction | 27.1 | 58.1
Statistical Analysis 1: Comparison: XEN-45 Gel Stent vs Trabeculectomy; Percentage of Participants Achieving Specific Percentage IOP Lower Targets From Baseline at Month 12 With Medication-free Eyes: ≥ 25% IOP Reduction; Test type: Other — No formal hypothesis was planned. P-value for treatment differences was provided for reference; p = 0.464, Fisher Exact; Percentage Difference = -9.6, 95% CI 2-sided [-31.0 to 12.1]
Statistical Analysis 2: Comparison: XEN-45 Gel Stent vs Trabeculectomy; Percentage of Participants Achieving Specific Percentage IOP Lower Targets From Baseline at Month 12 With Medication-free Eyes: ≥30% IOP Reduction; Test type: Other — No formal hypothesis was planned. P-value for treatment differences was provided for reference; p = 0.069, Fisher Exact; Percentage Difference = -19.8, 95% CI 2-sided [-40.6 to 2.1]
Statistical Analysis 3: Comparison: XEN-45 Gel Stent vs Trabeculectomy; Percentage of Participants Achieving Specific Percentage IOP Lower Targets From Baseline at Month 12 With Medication-free Eyes: ≥35% IOP Reduction; Test type: Other — No formal hypothesis was planned. P-value for treatment differences was provided for reference; p = 0.023, Fisher Exact; Percentage Difference = -26.6, 95% CI 2-sided [-46.9 to -4.7]
Statistical Analysis 4: Comparison: XEN-45 Gel Stent vs Trabeculectomy; Percentage of Participants Achieving Specific Percentage IOP Lower Targets From Baseline at Month 12 With Medication-free Eyes: ≥40% IOP Reduction; Test type: Other — No formal hypothesis was planned. P-value for treatment differences was provided for reference; p = 0.046, Fisher Exact; Percentage Difference = -23.7, 95% CI 2-sided [-43.9 to -1.6]
Statistical Analysis 5: Comparison: XEN-45 Gel Stent vs Trabeculectomy; Percentage of Participants Achieving Specific Percentage IOP Lower Targets From Baseline at Month 12 With Medication-free Eyes: ≥45% IOP Reduction; Test type: Other — No formal hypothesis was planned. P-value for treatment differences was provided for reference; p = 0.014, Fisher Exact; Percentage Difference = -27.6, 95% CI 2-sided [-47.6 to -5.9]
Statistical Analysis 6: Comparison: XEN-45 Gel Stent vs Trabeculectomy; Percentage of Participants Achieving Specific Percentage IOP Lower Targets From Baseline at Month 12 With Medication-free Eyes: ≥50% IOP Reduction; Test type: Other — No formal hypothesis was planned. P-value for treatment differences was provided for reference; p = 0.006, Fisher Exact; Percentage Difference = -30.9, 95% CI 2-sided [-50.8 to -9.5]

22. Secondary Outcome: Percentage of Participants With Intraoperative Adjunctive Antifibrotic Therapy Use
Description: Antifibrotic use included MMC which was standardized for both groups and administered according to physician training and practice.
Time Frame: Month 12
Population: Safety Population included all enrolled participants that have undergone study glaucoma surgery.
Measure: Number; unit: percentage of participants
Arm/Group | XEN-45 Gel Stent | Trabeculectomy
Number analyzed (Participants) | 95 | 44
percentage of participants | 98.9 | 97.7

23. Secondary Outcome: Percentage of Participants With Intraoperative Adjunctive Antifibrotic Therapy Based on Time of Administration
Description: Antifibrotic use included MMC which was standardized for both groups and administered according to physician training and practice. The time of administration was classified into two categories as: Before Procedure and After Procedure.
Time Frame: Month 12
Population: Safety Population included all enrolled participants that have undergone study glaucoma surgery.
Measure: Number; unit: percentage of participants
Arm/Group | XEN-45 Gel Stent | Trabeculectomy
Number analyzed (Participants) | 95 | 44
percentage of participants
  Before Procedure | 37.9 | 56.8
  After Procedure | 61.1 | 40.9

24. Secondary Outcome: Percentage of Participants With Different Modes of Administration of Intraoperative Adjunctive Antifibrotic Therapy
Description: Antifibrotic use included MMC which was standardized for both groups and administered according to physician training and practice. The mode of administration was classified into two categories as: Injection and Other. Other includes all other modes of administration apart from injection.
Time Frame: Month 12
Population: Safety Population included all enrolled participants that have undergone study glaucoma surgery.
Measure: Number; unit: percentage of participants
Arm/Group | XEN-45 Gel Stent | Trabeculectomy
Number analyzed (Participants) | 95 | 44
percentage of participants
  Injection | 98.9 | 84.1
  Other | 0 | 13.6

25. Secondary Outcome: Percentage of Participants With Different Volumes of Intraoperative Adjunctive Antifibrotic Therapy
Description: Antifibrotic use included MMC which was standardized for both groups and administered according to physician training and practice. The volume of administration measured in milliliters (mL) was classified into three categories as: 0.1, 0.2, and Other. Other includes all other volumes apart from 0.1 and 0.2.
Time Frame: Month 12
Population: Safety Population included all enrolled participants that have undergone study glaucoma surgery.
Measure: Number; unit: percentage of participants
Arm/Group | XEN-45 Gel Stent | Trabeculectomy
Number analyzed (Participants) | 95 | 44
percentage of participants
  0.1 | 50.5 | 34.1
  0.2 | 47.4 | 56.8
  Other | 1.1 | 2.3

26. Secondary Outcome: Percentage of Participants With Different Concentrations for Intraoperative Adjunctive Antifibrotic Therapy
Description: Antifibrotic use included MMC which was standardized for both groups and administered according to physician training and practice. The concentration of administration measured in milligram per milliliter (mg/mL) was classified into three categories as: 0.2, 0.4, and Other. Other includes all other concentrations apart from 0.2 and 0.4.
Time Frame: Month 12
Population: Safety Population included all enrolled participants that have undergone study glaucoma surgery.
Measure: Number; unit: percentage of participants
Arm/Group | XEN-45 Gel Stent | Trabeculectomy
Number analyzed (Participants) | 95 | 44
percentage of participants
  0.2 | 34.7 | 36.4
  0.4 | 64.2 | 56.8
  Other | 0 | 0

27. Secondary Outcome: Percentage of Participants With Different Absolute Dose for Intraoperative Adjunctive Antifibrotic Therapy
Description: Antifibrotic use included MMC which was standardized for both groups and administered according to physician training and practice. The absolute dose of administration measured in microgram per milliliter (µg/mL) was classified into two categories as: 40, and Other. Other includes all other concentrations apart from 40.
Time Frame: Month 12
Population: Safety Population included all enrolled participants that have undergone study glaucoma surgery.
Measure: Number; unit: percentage of participants
Arm/Group | XEN-45 Gel Stent | Trabeculectomy
Number analyzed (Participants) | 95 | 44
percentage of participants
  40 | 97.9 | 93.2
  Other | 1.1 | 0

28. Secondary Outcome: Mean Change From Baseline in Best Corrected Visual Acuity (BCVA) With Current Glasses
Description: BCVA was performed using a Snellen eye chart with glasses, and the BCVA data collected in the visual acuity electronic case report form (eCRF) page was analyzed. The number of lines read correctly was assessed as the line change from baseline at each follow-up evaluation and were log transformed. A logMAR value of 0 equates to 20/20 Snellen visual acuity (normal distance eyesight), with a lower and negative logMAR value indicating better visual acuity.
Time Frame: Baseline and Day 1, Weeks 1 and 2, and Months 1, 3, 6, 9, and 12
Population: ITT Population included all enrolled eyes/participants that were randomized to and received study glaucoma surgery (XEN-45 or trabeculectomy). Analyses were based on the randomized surgery. Number analyzed is the number of participants with data available for analysis at the given timepoint.
Measure: Least Squares Mean (Standard Error); unit: Log10 (Lines)
Arm/Group | XEN-45 Gel Stent | Trabeculectomy
Number analyzed (Participants) | 95 | 44
Log10 (Lines)
  Change From Baseline at Day 1: number analyzed (Participants) | 90 | 43
  Change From Baseline at Day 1 | -1.4 (0.20) | -2.5 (0.29)
  Change From Baseline at Week 1: number analyzed (Participants) | 87 | 42
  Change From Baseline at Week 1 | -1.2 (0.20) | -2.4 (0.29)
  Change From Baseline at Week 2: number analyzed (Participants) | 90 | 42
  Change From Baseline at Week 2 | -1.1 (0.20) | -1.6 (0.29)
  Change From Baseline at Month 1: number analyzed (Participants) | 92 | 39
  Change From Baseline at Month 1 | -0.6 (0.20) | -1.1 (0.30)
  Change From Baseline at Month 3: number analyzed (Participants) | 87 | 39
  Change From Baseline at Month 3 | -0.4 (0.20) | -0.5 (0.30)
  Change From Baseline at Month 6: number analyzed (Participants) | 81 | 40
  Change From Baseline at Month 6 | -0.4 (0.21) | -0.4 (0.30)
  Change From Baseline at Month 9: number analyzed (Participants) | 81 | 39
  Change From Baseline at Month 9 | -0.4 (0.21) | -1.0 (0.30)
  Change From Baseline at Month 12: number analyzed (Participants) | 74 | 36
  Change From Baseline at Month 12 | -0.1 (0.21) | -0.8 (0.31)
Statistical Analysis 1: Comparison: XEN-45 Gel Stent vs Trabeculectomy; Mean Change From Baseline in Best Corrected Visual Acuity (BCVA) With Current Glasses: Day 1; Test type: Other — No formal hypothesis was planned. P-value for treatment differences was provided for reference; p = 0.004, Mixed Model for Repeated Measures; MMRM model with treatment and time as the factors, treatment by time interaction and baseline as the covariate variables were used for analysis; Least Square Mean Difference = 1.0, 95% CI 2-sided [0.33 to 1.72], Standard Error of Mean 0.35
Statistical Analysis 2: Comparison: XEN-45 Gel Stent vs Trabeculectomy; Mean Change From Baseline in Best Corrected Visual Acuity (BCVA) With Current Glasses:Week 1; Test type: Other — No formal hypothesis was planned. P-value for treatment differences was provided for reference; p = 0.001, Mixed Model for Repeated Measures — [p-value comment as in outcome 3, analysis 2]; Least Square Mean Difference = 1.2, 95% CI 2-sided [0.47 to 1.88], Standard Error of Mean 0.36
Statistical Analysis 3: Comparison: XEN-45 Gel Stent vs Trabeculectomy; Mean Change From Baseline in Best Corrected Visual Acuity (BCVA) With Current Glasses:Week 2; Test type: Other — No formal hypothesis was planned. P-value for treatment differences was provided for reference; p = 0.162, Mixed Model for Repeated Measures — [p-value comment as in outcome 3, analysis 2]; Least Square Mean Difference = 0.5, 95% CI 2-sided [-0.20 to 1.20], Standard Error of Mean 0.36
Statistical Analysis 4: Comparison: XEN-45 Gel Stent vs Trabeculectomy; Mean Change From Baseline in Best Corrected Visual Acuity (BCVA) With Current Glasses:Month 1; Test type: Other — No formal hypothesis was planned. P-value for treatment differences was provided for reference; p = 0.185, Mixed Model for Repeated Measures — [p-value comment as in outcome 3, analysis 2]; Least Square Mean Difference = 0.5, 95% CI 2-sided [-0.23 to 1.19], Standard Error of Mean 0.36
Statistical Analysis 5: Comparison: XEN-45 Gel Stent vs Trabeculectomy; Mean Change From Baseline in Best Corrected Visual Acuity (BCVA) With Current Glasses:Month 3; Test type: Other — No formal hypothesis was planned. P-value for treatment differences was provided for reference; p = 0.846, Mixed Model for Repeated Measures — [p-value comment as in outcome 3, analysis 2]; Least Square Mean Difference = 0.1, 95% CI 2-sided [-0.64 to 0.79], Standard Error of Mean 0.36
Statistical Analysis 6: Comparison: XEN-45 Gel Stent vs Trabeculectomy; Mean Change From Baseline in Best Corrected Visual Acuity (BCVA) With Current Glasses:Month 6; Test type: Other — No formal hypothesis was planned. P-value for treatment differences was provided for reference; p = 0.965, Mixed Model for Repeated Measures — [p-value comment as in outcome 3, analysis 2]; Least Square Mean Difference = 0.0, 95% CI 2-sided [-0.73 to 0.70], Standard Error of Mean 0.36
Statistical Analysis 7: Comparison: XEN-45 Gel Stent vs Trabeculectomy; Mean Change From Baseline in Best Corrected Visual Acuity (BCVA) With Current Glasses:Month 9; Test type: Other — No formal hypothesis was planned. P-value for treatment differences was provided for reference; p = 0.096, Mixed Model for Repeated Measures — [p-value comment as in outcome 3, analysis 2]; Least Square Mean Difference = 0.6, 95% CI 2-sided [-0.11 to 1.33], Standard Error of Mean 0.37
Statistical Analysis 8: Comparison: XEN-45 Gel Stent vs Trabeculectomy; Mean Change From Baseline in Best Corrected Visual Acuity (BCVA) With Current Glasses:Month 12; Test type: Other — No formal hypothesis was planned. P-value for treatment differences was provided for reference; p = 0.063, Mixed Model for Repeated Measures — [p-value comment as in outcome 3, analysis 2]; Least Square Mean Difference = 0.7, 95% CI 2-sided [-0.04 to 1.43], Standard Error of Mean 0.37

29. Secondary Outcome: Mean Change From Baseline in Manifest Refraction - Mean Visual Acuity Using Snellen Eye Chart in LogMAR Scale
Description: Manifest Refraction - Mean Visual Acuity was performed using a Snellen eye chart with glasses. The line change from baseline at each follow-up evaluation in logarithm of the minimum angle of resolution (logMAR) was calculated. A logMAR value of 0 equates to 20/20 Snellen visual acuity (normal distance eyesight), with a lower logMAR value indicating better visual acuity.
Time Frame: Baseline (Preoperative) and postoperative Months 1, 3, 6, and 12
Population: as for outcome 28
Measure: Least Squares Mean (Standard Error); unit: logMAR
Arm/Group | XEN-45 Gel Stent | Trabeculectomy
Number analyzed (Participants) | 95 | 44
logMAR
  Change From Baseline at Month 1: number analyzed (Participants) | 77 | 40
  Change From Baseline at Month 1 | 0.05 (0.015) | 0.10 (0.022)
  Change From Baseline at Month 3: number analyzed (Participants) | 70 | 37
  Change From Baseline at Month 3 | 0.04 (0.016) | 0.05 (0.022)
  Change From Baseline at Month 6: number analyzed (Participants) | 69 | 37
  Change From Baseline at Month 6 | 0.04 (0.016) | 0.04 (0.022)
  Change From Baseline at Month 12: number analyzed (Participants) | 67 | 35
  Change From Baseline at Month 12 | 0.01 (0.016) | 0.07 (0.022)
Statistical Analysis 1: Comparison: XEN-45 Gel Stent vs Trabeculectomy; Mean Change From Baseline in Manifest Refraction - Mean Visual Acuity Using Snellen in LogMAR Scale: Month 1; Test type: Other — No formal hypothesis was planned. P-value for treatment differences was provided for reference; p = 0.048, Mixed Model for Repeated Measures; Least Square Mean Difference = -0.05, 95% CI 2-sided [-0.105 to 0.000], Standard Error of Mean 0.027
Statistical Analysis 2: Comparison: XEN-45 Gel Stent vs Trabeculectomy; Mean Change From Baseline in Manifest Refraction - Mean Visual Acuity Using Snellen in LogMAR Scale: Month 3; Test type: Other — No formal hypothesis was planned. P-value for treatment differences was provided for reference; p = 0.742, Mixed Model for Repeated Measures; Least Square Mean Difference = -0.01, 95% CI 2-sided [-0.062 to 0.045], Standard Error of Mean 0.027
Statistical Analysis 3: Comparison: XEN-45 Gel Stent vs Trabeculectomy; Mean Change From Baseline in Manifest Refraction - Mean Visual Acuity Using Snellen in LogMAR Scale: Month 6; Test type: Other — No formal hypothesis was planned. P-value for treatment differences was provided for reference; p = 0.925, Mixed Model for Repeated Measures; Least Square Mean Difference = 0.00, 95% CI 2-sided [-0.056 to 0.051], Standard Error of Mean 0.027
Statistical Analysis 4: Comparison: XEN-45 Gel Stent vs Trabeculectomy; Mean Change From Baseline in Manifest Refraction - Mean Visual Acuity Using Snellen in LogMAR Scale: Month 12; Test type: Other — No formal hypothesis was planned. P-value for treatment differences was provided for reference; p = 0.021, Mixed Model for Repeated Measures; Least Square Mean Difference = -0.06, 95% CI 2-sided [-0.118 to -0.010], Standard Error of Mean 0.028

30. Secondary Outcome: Mean Surgically Induced Astigmatism - Autorefractor Reading
Time Frame: Month 12
Population: No data is reported due to inaccuracy of the results (autorefractor reading errors).
Arm/Group | XEN-45 Gel Stent | Trabeculectomy
Number analyzed (Participants) | 0 | 0

31. Secondary Outcome: Mean Change From Baseline in Surgically Induced Astigmatism - Autorefractor Reading
Time Frame: Baseline (Preoperative) and Month 12
Population: No data is reported due to inaccuracy of the results (autorefractor reading errors).
Arm/Group | XEN-45 Gel Stent | Trabeculectomy
Number analyzed (Participants) | 0 | 0

32. Secondary Outcome: Mean Change From Baseline in Surgically Induced Astigmatism - Topography at Selected Sites
Time Frame: Baseline (Preoperative), Week 1, and Months 1 and 12
Population: ITT Population included all enrolled eyes/participants that were randomized to and received study glaucoma surgery (XEN-45 or trabeculectomy). Analyses were based on the randomized surgery. Overall Number of Participants Analyzed is the number of participants with data available for analyses at Baseline. Number Analyzed is the number of participants with data available for analyses at Baseline and the given timepoint.
Measure: Least Squares Mean (Standard Error); unit: diopters
Arm/Group | XEN-45 Gel Stent | Trabeculectomy
Number analyzed (Participants) | 23 | 12
diopters
  Change From Baseline at Week 1: number analyzed (Participants) | 20 | 10
  Change From Baseline at Week 1 | 0.057 (0.1861) | 0.619 (0.2639)
  Change From Baseline at Month 1: number analyzed (Participants) | 18 | 9
  Change From Baseline at Month 1 | 0.187 (0.1931) | 0.326 (0.2741)
  Change From Baseline at Month 12: number analyzed (Participants) | 17 | 8
  Change From Baseline at Month 12 | 0.106 (0.1976) | 0.558 (0.2860)
Statistical Analysis 1: Comparison: XEN-45 Gel Stent vs Trabeculectomy; Mean Change from Baseline in Surgically Induced Astigmatism - Topography at Selected Sites at Week 1; Test type: Other — No formal hypothesis was planned. P-value for treatment differences was provided for reference; p = 0.087, Mixed Model for Repeated Measures; Least Square Mean Difference = -0.562, 95% CI 2-sided [-1.2082 to 0.0851], Standard Error of Mean 0.3231
Statistical Analysis 2: Comparison: XEN-45 Gel Stent vs Trabeculectomy; Mean Change from Baseline in Surgically Induced Astigmatism - Topography at Selected Sites at Month 1; Test type: Other — No formal hypothesis was planned. P-value for treatment differences was provided for reference; p = 0.682, Mixed Model for Repeated Measures; Least Square Mean Difference = -0.138, 95% CI 2-sided [-0.8090 to 0.5324], Standard Error of Mean 0.3355
Statistical Analysis 3: Comparison: XEN-45 Gel Stent vs Trabeculectomy; Mean Change from Baseline in Surgically Induced Astigmatism - Topography at Selected Sites at Month 12; Test type: Other — No formal hypothesis was planned. P-value for treatment differences was provided for reference; p = 0.199, Mixed Model for Repeated Measures; Least Square Mean Difference = -0.452, 95% CI 2-sided [-1.1483 to 0.2434], Standard Error of Mean 0.3484

33. Secondary Outcome: Mean Change From Baseline in Optical Biometry - Anterior Chamber Depth
Time Frame: Baseline, Day 1 and Week 2
Population: as for outcome 32
Measure: Least Squares Mean (Standard Error); unit: millimeter
Arm/Group | XEN-45 Gel Stent | Trabeculectomy
Number analyzed (Participants) | 21 | 10
millimeter
  Change from Baseline at Day 1: number analyzed (Participants) | 14 | 10
  Change from Baseline at Day 1 | -0.183 (0.1295) | -0.182 (0.1553)
  Change from Baseline at Week 2: number analyzed (Participants) | 17 | 8
  Change from Baseline at Week 2 | -0.206 (0.1195) | -0.427 (0.1732)
Statistical Analysis 1: Comparison: XEN-45 Gel Stent vs Trabeculectomy; Mean Change in Optical Biometry - Anterior Chamber Depth at Day 1; Test type: Other — No formal hypothesis was planned. P-value for treatment differences was provided for reference; p = 0.997, Mixed Model for Repeated Measures; Least Square Mean Difference = -0.001, 95% CI 2-sided [-0.4103 to 0.4086], Standard Error of Mean 0.2026
Statistical Analysis 2: Comparison: XEN-45 Gel Stent vs Trabeculectomy; Mean Change in Optical Biometry - Anterior Chamber Depth at Week 2; Test type: Other — No formal hypothesis was planned. P-value for treatment differences was provided for reference; p = 0.302, Mixed Model for Repeated Measures; Least Square Mean Difference = 0.222, 95% CI 2-sided [-0.2068 to 0.6506], Standard Error of Mean 0.2124

34. Secondary Outcome: Mean Change in From Baseline Optical Biometry - Keratometry (K)1, K2, Delta D
Description: The keratometric values for keratometry (K) measured in 2 meridians (i.e., flat keratometry [K1] and steep keratometry [K2]) along with Delta (D) were determined.
Time Frame: Baseline, Day 1 and Week 2
Population: as for outcome 32
Measure: Least Squares Mean (Standard Error); unit: diopter
Arm/Group | XEN-45 Gel Stent | Trabeculectomy
Number analyzed (Participants) | 21 | 12
diopter
  K1, Change from Baseline at Day 1: number analyzed (Participants) | 14 | 11
  K1, Change from Baseline at Day 1 | -0.103 (0.2195) | -0.446 (0.2512)
  K1, Change from Baseline at Week 2: number analyzed (Participants) | 18 | 10
  K1, Change from Baseline at Week 2 | 0.156 (0.1973) | -0.105 (0.2618)
  K2, Change from Baseline at Day 1: number analyzed (Participants) | 14 | 11
  K2, Change from Baseline at Day 1 | 0.373 (0.2947) | 0.783 (0.3342)
  K2, Change from Baseline at Week 2: number analyzed (Participants) | 18 | 10
  K2, Change from Baseline at Week 2 | 0.152 (0.2626) | 0.640 (0.3499)
  Delta D, Change from Baseline at Day 1: number analyzed (Participants) | 14 | 11
  Delta D, Change from Baseline at Day 1 | 0.514 (0.2967) | 1.279 (0.3372)
  Delta D, Change from Baseline at Week 2: number analyzed (Participants) | 18 | 10
  Delta D, Change from Baseline at Week 2 | 0.087 (0.2636) | 0.664 (0.3527)
Statistical Analysis 1: Comparison: XEN-45 Gel Stent vs Trabeculectomy; Mean Change in from Baseline Optical Biometry - K1 at Day 1; Test type: Other — No formal hypothesis was planned. P-value for treatment differences was provided for reference; p = 0.309, Mixed Model for Repeated Measures; Least Square Mean Difference = 0.343, 95% CI 2-sided [-0.3289 to 1.0154], Standard Error of Mean 0.3336
Statistical Analysis 2: Comparison: XEN-45 Gel Stent vs Trabeculectomy; Mean Change in from Baseline Optical Biometry - K1 at Week 2; Test type: Other — No formal hypothesis was planned. P-value for treatment differences was provided for reference; p = 0.430, Mixed Model for Repeated Measures; Least Square Mean Difference = 0.261, 95% CI 2-sided [-0.3993 to 0.9220], Standard Error of Mean 0.3278
Statistical Analysis 3: Comparison: XEN-45 Gel Stent vs Trabeculectomy; Mean Change in from Baseline Optical Biometry - K2 at Day 1; Test type: Other — No formal hypothesis was planned. P-value for treatment differences was provided for reference; p = 0.363, Mixed Model for Repeated Measures; Least Square Mean Difference = -0.409, 95% CI 2-sided [-1.3071 to 0.4882], Standard Error of Mean 0.4457
Statistical Analysis 4: Comparison: XEN-45 Gel Stent vs Trabeculectomy; Mean Change in from Baseline Optical Biometry - K2 at Week 2; Test type: Other — No formal hypothesis was planned. P-value for treatment differences was provided for reference; p = 0.272, Mixed Model for Repeated Measures; Least Square Mean Difference = -0.488, 95% CI 2-sided [-1.3709 to 0.3954], Standard Error of Mean 0.4383
Statistical Analysis 5: Comparison: XEN-45 Gel Stent vs Trabeculectomy; Mean Change in from Baseline Optical Biometry - Delta D at Day 1; Test type: Other — No formal hypothesis was planned. P-value for treatment differences was provided for reference; p = 0.096, Mixed Model for Repeated Measures; Least Square Mean Difference = -0.765, 95% CI 2-sided [-1.6722 to 0.1420], Standard Error of Mean 0.4502
Statistical Analysis 6: Comparison: XEN-45 Gel Stent vs Trabeculectomy; Mean Change in from Baseline Optical Biometry - Delta D at Week 2; Test type: Other — No formal hypothesis was planned. P-value for treatment differences was provided for reference; p = 0.198, Mixed Model for Repeated Measures; Least Square Mean Difference = -0.576, 95% CI 2-sided [-1.4655 to 0.3129], Standard Error of Mean 0.4411

35. Secondary Outcome: Bleb Morphology - Anterior Segment Optical Coherence Tomography (AS-OCT) at Selected Sites
Time Frame: Up to Month 12
Population: No tabular data was collected. Photographs were taken at select sites to be used for publication purposes.
Arm/Group | XEN-45 Gel Stent | Trabeculectomy
Number analyzed (Participants) | 0 | 0

36. Secondary Outcome: Bleb Morphology - Slit Lamp Photography at Selected Sites
Time Frame: Up to Month 12
Population: No tabular data was collected. Photographs were taken at select sites to be used for publication purposes.
Arm/Group | XEN-45 Gel Stent | Trabeculectomy
Number analyzed (Participants) | 0 | 0

37. Secondary Outcome: Percentage of Participants With Clinical Hypotony
Description: Clinical hypotony was defined as vision reduction (2 lines or more) related to macular changes consistent with hypotony maculopathy (macular folds), optic disc edema, and/or serous choroidal detachments because of low IOP.
Time Frame: Month 12
Population: Safety Population included all enrolled participants that have undergone study glaucoma surgery.
Measure: Number; unit: percentage of participants
Arm/Group | XEN-45 Gel Stent | Trabeculectomy
Number analyzed (Participants) | 95 | 44
percentage of participants | 23.2 | 50.0

38. Secondary Outcome: Percentage of Eyes With IOP 6 mm Hg or Less at Any Time Point and Relevant Clinical Assessment
Description: Eyes with IOP 6 mm Hg or less at any time point and relevant clinical assessment (vision reduction [2 lines or more] related to macular changes consistent with hypotony maculopathy [macular folds], optic disc edema, anterior chamber status, and/or serous choroidal detachments because of low IOP) of these eyes at those time points were assessed. Only data from study eyes are included. The worse eye was selected as the study eye if both eyes met the inclusion criteria. The worse eye was defined using the visual field MD at Baseline, with the worse eye having the most negative MD. In cases where the MD was the same in both eyes to two decimal places, the worse eye was defined as the eye with the higher IOP.
Time Frame: Up to Month 12
Population: Safety Population included all enrolled participants/eyes that have undergone study glaucoma surgery.
Measure: Number; unit: percentage of eyes
Units Other Than Participants: eyes
Arm/Group | XEN-45 Gel Stent | Trabeculectomy
Number analyzed (Participants) | 95 | 44
Number analyzed (eyes) | 95 | 44
percentage of eyes | 13.7 | 29.5

39. Secondary Outcome: Percentage of Participants With Specific Intraoperative Adverse Events of Special Interest (AESIs)
Description: An adverse event(AE)is any untoward medical occurrence in a clinical investigation participant administered drug; it does not necessarily have to have a causal relationship with the treatment. Intraoperative AESIs included- Detached Descemet's membrane,iris damage,lens contact,vitreous bulge or loss,anterior chamber bleeding,retrobulbar hemorrhage,conjunctival perforation,conjunctival or scleral flap tearing,shallow anterior chamber with peripheral iridocorneal touch,flat anterior chamber with iridocorneal touch extending to the pupil,device malfunction identified prior to implantation,and choroidal hemorrhage of effusion. Only categories with at least one participant with event in the study eye are reported. The worse eye was selected as the study eye if both eyes met inclusion criteria. The worse eye was defined using visual field MD at Baseline, with the worse eye having the most negative MD. If MD was same in both eyes to two decimal places, the worse eye=eye with higher IOP.
Time Frame: Median follow-up of 366.0 days
Population: Safety Population included all enrolled participants that have undergone study glaucoma surgery.
Measure: Number; unit: percentage of participants
Arm/Group | XEN-45 Gel Stent | Trabeculectomy
Number analyzed (Participants) | 95 | 44
percentage of participants
  Anterior Chamber Bleeding | 1.1 | 4.5
  Other | 1.1 | 2.3
  Conjunctival Buttonhole | 0.0 | 2.3
  Iris Damage | 0.0 | 2.3

40. Secondary Outcome: Percentage of Participants With Postoperative Treatment-Emergent Adverse Events of Special Interest (AESIs)
Description: AE=any untoward medical occurrence in a clinical investigation participant administered drug;it does not necessarily have to have a causal relationship with the treatment. TEAE is an AE either reported for the first time or worsening of a pre-existing event after first dose of study drug and within 30 days of the last administration of study drug. Postoperative AEs included but were not limited to: angle recession, anterior chamber changes, BCVA loss,bleb leak, blebitis, cataract, choroidal effusion, chronic pain, corneal edema, cyclodialysis, Dellen, device malfunction, endophthalmitis, fixed dilated pupil, hyphema, hypotony, implant issues, increase in corneal thickness/IOP, explant, iridodialysis, iritis, loss of eye, etc.Worse eye=eye if both eyes met inclusion criteria. Worse eye was defined using visual field MD at Baseline, with worse eye having the most negative MD. In cases where MD was the same in both eyes to two decimal places, worse eye was defined as eye with higher IOP.
Time Frame: Median follow-up of 366.0 days
Population: Safety Population included all enrolled participants that have undergone study glaucoma surgery.
Measure: Number; unit: percentage of participants
Arm/Group | XEN-45 Gel Stent | Trabeculectomy
Number analyzed (Participants) | 95 | 44
percentage of participants | 66.3 | 86.4

41. Secondary Outcome: Percentage of Participants With BCVA Worst Line Change From Baseline Across Follow-Up
Description: The categories = Worsening (<-2), No Change (≥-2 and ≥2), Improving (>2) and Missing were used for determining BCVA worst line change from Baseline. Only categories with at least one participant with event are reported.
Time Frame: Baseline up to Month 12
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | XEN-45 Gel Stent | Trabeculectomy
Number analyzed (Participants) | 95 | 44
percentage of participants
  Worsening | 36.84 | 56.82
  No Change | 63.16 | 40.91
  Missing | 0.0 | 2.27

42. Secondary Outcome: Pachymetry Based on Change From Baseline In Average Central Corneal Thickness
Description: Pachymetry was measured as average central corneal thickness (microns/micrometer) change from Baseline.
Time Frame: Baseline (Preoperative) and Month 12
Population: Safety Population included all enrolled participants that have undergone study glaucoma surgery. Overall number analyzed are the number of participants with data available for analyses.
Measure: Mean (Standard Deviation); unit: micrometer (µm)
Arm/Group | XEN-45 Gel Stent | Trabeculectomy
Number analyzed (Participants) | 64 | 30
micrometer (µm) | -2.0 (21.41) | 6.4 (12.44)

43. Secondary Outcome: Change From Baseline in Visual Field Examinations Analyzed by Machine Type
Description: All visual field examination data were collected and reported as mean deviation by Humphrey machine.
Time Frame: Baseline and Month 12
Population: as for outcome 42
Measure: Mean (Standard Deviation); unit: decibel (dB)
Arm/Group | XEN-45 Gel Stent | Trabeculectomy
Number analyzed (Participants) | 68 | 34
decibel (dB) | -0.051 (4.5578) | -0.356 (3.0171)

44. Secondary Outcome: Percentage of Participants With at Least One Adverse Event (AE), Serious Adverse Events (SAEs), Adverse Device Effects (ADEs) and Serious ADEs (SADEs)
Description: AE=any untoward medical occurrence in a clinical investigation participant administered drug; it does not necessarily have to have a causal relationship with the treatment. An SAE was defined as any untoward medical occurrence that: 1) results in death, 2) is life-threatening, 3) requires inpatient hospitalization or prolongation of existing hospitalization, 4) results in persistent or significant disability/incapacity, 5) leads to a congenital anomaly/birth defect in the offspring of the participant or 6) is a medically important event that satisfies any of the following: a) May require intervention to prevent items 1 through 5 above. b) May expose the participant to danger, even though the event is not immediately life threatening or fatal or does not result in hospitalization. ADEs and SADEs are AEs and SAEs that are caused by the device
Time Frame: Median follow-up of 366.0 days
Population: Safety Population included all enrolled participants that have undergone study glaucoma surgery.
Measure: Number; unit: percentage of participants
Arm/Group | XEN-45 Gel Stent | Trabeculectomy
Number analyzed (Participants) | 95 | 44
percentage of participants
  TEAEs | 74.7 | 93.2
  TESAEs | 9.5 | 4.5
  TEADEs | 0.0 | 0.0
  TESADEs | 0.0 | 0.0

45. Secondary Outcome: Patient-reported Outcomes (PRO): Change From Baseline in Symptom and Health Problem Checklist (SHPC-18) Scores
Description: The SHPC-18 is an 18-item questionnaire that asks participants being treated for glaucoma questions about eye symptoms or problems they may experience. There are two domains: Local Eye Symptoms (7 items) subscale score 0 to 700 divided by 7 and Visual Function Problem (11 items) subscale score 0 to 1100 divided by 11. The scores of each subscale ranges from from 0 (not at all) to 100 (a lot); higher scores indicate more bother. A frequency score was calculated by summing the individual response scores of each item, and ranges from 0 to 7 for Local Eye Symptom and from 0 to 11 for Visual Function. A total bothersome score for the SHPC-18 is calculated by summing all 18 items scores, resulting in a range from 0 to 1800, then dividing the sum by 18, to create a total bothersome score ranging from 0 (not at all) to 100 (a lot); higher scores indicate more bother. A negative change from Baseline for all scales and subscales indicates improvement.
Time Frame: Baseline (Preoperative) to Month 6
Population: as for outcome 7
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | XEN-45 Gel Stent | Trabeculectomy
Number analyzed (Participants) | 44 | 26
score on a scale
  Local Eye Symptoms Score | -3.328 (2.5560) | -0.297 (3.4928)
  Vision Function Problem Score | -3.064 (2.6759) | 7.443 (3.6965)
  Total Bothersome Score | -3.160 (2.3564) | 4.368 (3.2737)
  Local Eye Symptoms Frequency Score | -0.6 (0.25) | -0.1 (0.34)
  Vision Function Problem Frequency Score | -0.7 (0.37) | 1.0 (0.51)
Statistical Analysis 1: Comparison: XEN-45 Gel Stent vs Trabeculectomy; PRO: Change From Baseline in Symptom and Health Problem Checklist (SHPC-18)- Local Eye Symptoms Score; Test type: Other — No formal hypothesis was planned. P-value for treatment differences was provided for reference; p = 0.485, Mixed Model for Repeated Measures; Least Square Mean Difference = -3.031, 95% CI 2-sided [-11.5597 to 5.4973], Standard Error of Mean 4.3331
Statistical Analysis 2: Comparison: XEN-45 Gel Stent vs Trabeculectomy; PRO: Change From Baseline in Symptom and Health Problem Checklist (SHPC-18)- Vision Function Problem Score; Test type: Other — No formal hypothesis was planned. P-value for treatment differences was provided for reference; p = 0.022, Mixed Model for Repeated Measures; Least Square Mean Difference = -10.507, 95% CI 2-sided [-19.5000 to -1.5144], Standard Error of Mean 4.5666
Statistical Analysis 3: Comparison: XEN-45 Gel Stent vs Trabeculectomy; PRO: Change From Baseline in Symptom and Health Problem Checklist (SHPC-18)- Total Bothersome Score; Test type: Other — No formal hypothesis was planned. P-value for treatment differences was provided for reference; p = 0.064, Mixed Model for Repeated Measures; Least Square Mean Difference = -7.528, 95% CI 2-sided [-15.4841 to 0.4275], Standard Error of Mean 4.0382
Statistical Analysis 4: Comparison: XEN-45 Gel Stent vs Trabeculectomy; PRO: Change From Baseline in Symptom and Health Problem Checklist (SHPC-18)- Local Eye Symptoms Frequency Score; Test type: Other — No formal hypothesis was planned. P-value for treatment differences was provided for reference; p = 0.278, Mixed Model for Repeated Measures; Least Square Mean Difference = -0.5, 95% CI 2-sided [-1.28 to 0.37], Standard Error of Mean 0.42
Statistical Analysis 5: Comparison: XEN-45 Gel Stent vs Trabeculectomy; PRO: Change From Baseline in Symptom and Health Problem Checklist (SHPC-18)- Vision Function Problem Frequency Score; Test type: Other — No formal hypothesis was planned. P-value for treatment differences was provided for reference; p = 0.007, Mixed Model for Repeated Measures; Least Square Mean Difference = -1.7, 95% CI 2-sided [-2.96 to -0.47], Standard Error of Mean 0.63

46. Secondary Outcome: PRO: Percentage of Participants With Post-Surgical Resumption of Activities and Daily Routine
Description: Participants answered the question, "Since your glaucoma surgery, would you consider that you have resumed your usual activities and daily routine?" using the following categories: Not at all, Somewhat, Moderately so, Mostly, Completely.
Time Frame: Month 3
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | XEN-45 Gel Stent | Trabeculectomy
Number analyzed (Participants) | 95 | 44
percentage of participants
  Not at all | 1.1 | 2.3
  Somewhat | 4.2 | 9.1
  Moderately so | 4.2 | 4.5
  Mostly | 6.3 | 20.5
  Completely | 41.1 | 31.8
  Missing | 43.2 | 31.8
Statistical Analysis 1: Comparison: XEN-45 Gel Stent vs Trabeculectomy; PRO: Percentage of Participants With Post-Surgical Resumption of Activities and Daily Routine- Not at all; Test type: Other — No formal hypothesis was planned. P-value for treatment differences was provided for reference; p = 0.534, Fisher Exact
Statistical Analysis 2: Comparison: XEN-45 Gel Stent vs Trabeculectomy; PRO: Percentage of Participants With Post-Surgical Resumption of Activities and Daily Routine- Somewhat; Test type: Other — No formal hypothesis was planned. P-value for treatment differences was provided for reference; p = 0.263, Fisher Exact
Statistical Analysis 3: Comparison: XEN-45 Gel Stent vs Trabeculectomy; PRO: Percentage of Participants With Post-Surgical Resumption of Activities and Daily Routine- Moderately so; Test type: Other — No formal hypothesis was planned. P-value for treatment differences was provided for reference; p = 1.000, Fisher Exact
Statistical Analysis 4: Comparison: XEN-45 Gel Stent vs Trabeculectomy; PRO: Percentage of Participants With Post-Surgical Resumption of Activities and Daily Routine- Mostly; Test type: Other — No formal hypothesis was planned. P-value for treatment differences was provided for reference; p = 0.018, Fisher Exact
Statistical Analysis 5: Comparison: XEN-45 Gel Stent vs Trabeculectomy; PRO: Percentage of Participants With Post-Surgical Resumption of Activities and Daily Routine- Completely; Test type: Other — No formal hypothesis was planned. P-value for treatment differences was provided for reference; p = 0.350, Fisher Exact
Statistical Analysis 6: Comparison: XEN-45 Gel Stent vs Trabeculectomy; PRO: Percentage of Participants With Post-Surgical Resumption of Activities and Daily Routine- Missing; Test type: Other — No formal hypothesis was planned. P-value for treatment differences was provided for reference; p = 0.264, Fisher Exact

47. Secondary Outcome: PRO: Percent Change From Baseline in Work Productivity and Activity Impairment (WPAI): Percent Overall Work Impairment Due to Health
Description: WPAI-General Health (GH) is 6-question participant rated questionnaire to determine the amount of absenteeism, presenteeism, work productivity loss and daily activity impairment attributable to general health. It yields 5 sub-scores: hours actually worked, work time missed due to health impairment while working, impairment while working due to health, overall work impairment due to health, activity impairment due to health. These sub-scores are transformed to impairment percentages (range from 0 to 100), with higher numbers indicating greater impairment and less productivity. A negative change from Baseline indicates improvement.
Time Frame: Baseline (Preoperative) and Month 12
Population: ITT Population included all enrolled eyes/participants that were randomized to and received study glaucoma surgery (XEN-45 or trabeculectomy). Analyses were based on the randomized surgery. Overall Number of Participants Analyzed is the number of participants with data available for analysis at the given timepoint.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | XEN-45 Gel Stent | Trabeculectomy
Number analyzed (Participants) | 5 | 7
percent change | -0.994 (12.4333) | 7.309 (10.3287)
Statistical Analysis 1: Comparison: XEN-45 Gel Stent vs Trabeculectomy; PRO: Percent Change From Baseline in Work Productivity and Activity Impairment- Percent Overall Work Impairment Due to Health; Test type: Other — No formal hypothesis was planned. P-value for treatment differences was provided for reference; p = 0.610, Mixed Model for Repeated Measures; Least Square Mean Difference = -8.303, 95% CI 2-sided [-40.8681 to 24.2624], Standard Error of Mean 16.1445

48. Secondary Outcome: PRO: Percent Change From Baseline in WPAI: Percent Activity Impairment Due to Health
Description: as for outcome 47
Time Frame: Baseline (Preoperative) and Month 12
Population: as for outcome 47
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | XEN-45 Gel Stent | Trabeculectomy
Number analyzed (Participants) | 30 | 19
percent change | -3.1 (5.18) | 10.8 (6.53)
Statistical Analysis 1: Comparison: XEN-45 Gel Stent vs Trabeculectomy; PRO: Percent Change From Baseline in Work Productivity and Activity Impairment-Percent Activity Impairment Due to Health; Test type: Other — No formal hypothesis was planned. P-value for treatment differences was provided for reference; p = 0.097, Mixed Model for Repeated Measures; Least Square Mean Difference = -13.9, 95% CI 2-sided [-30.32 to 2.52], Standard Error of Mean 8.33

ADVERSE EVENTS:
Time Frame: Median follow-up of 366.0 days
Description: All-Cause Mortality: Enrolled Population included all participants with study eyes for which participants had signed the informed consent form (ICF). SAEs and Other AEs: Safety Population included all enrolled participants with study eyes that have undergone study glaucoma surgery.
Arm/Group | XEN-45 Gel Stent | Trabeculectomy
All-Cause Mortality (participants affected / at risk) | 3/107 | 1/51
Serious Adverse Events (participants affected / at risk) | 9/95 | 2/44
Other Adverse Events (participants affected / at risk) | 59/95 | 38/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | XEN-45 Gel Stent (N=95) | Trabeculectomy (N=44)
CARDIAC ARREST (Cardiac disorders) | 1 (1) | 0 (0)
VISUAL ACUITY REDUCED (Eye disorders) | 1 (1) | 0 (0)
CORONA VIRUS INFECTION (Infections and infestations) | 2 (2) | 0 (0)
ENDOPHTHALMITIS (Infections and infestations) | 1 (1) | 0 (0)
PERIORBITAL CELLULITIS (Infections and infestations) | 1 (1) | 0 (0)
PNEUMONIA (Infections and infestations) | 1 (1) | 0 (0)
SEPSIS (Infections and infestations) | 1 (1) | 0 (0)
FALL (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
INTRAOCULAR PRESSURE INCREASED (Investigations) | 1 (1) | 0 (0)
PARKINSON'S DISEASE (Nervous system disorders) | 1 (1) | 0 (0)
DEVICE EXTRUSION (Product Issues) | 1 (1) | 0 (0)
ACUTE RESPIRATORY DISTRESS SYNDROME (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | XEN-45 Gel Stent (N=95) | Trabeculectomy (N=44)
CHOROIDAL EFFUSION (Eye disorders) | 2 (2) | 4 (5)
DRY EYE (Eye disorders) | 3 (3) | 3 (3)
GLAUCOMA (Eye disorders) | 0 (0) | 3 (3)
HYPOTONY OF EYE (Eye disorders) | 22 (24) | 22 (32)
PUNCTATE KERATITIS (Eye disorders) | 2 (2) | 3 (3)
VISUAL ACUITY REDUCED (Eye disorders) | 36 (59) | 24 (39)
CONJUNCTIVAL FILTERING BLEB LEAK (Injury, poisoning and procedural complications) | 0 (0) | 7 (9)
HYPHAEMA (Injury, poisoning and procedural complications) | 6 (6) | 3 (3)
INTRAOCULAR PRESSURE INCREASED (Investigations) | 19 (23) | 5 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2019-03-21): https://cdn.clinicaltrials.gov/large-docs/85/NCT03654885/Prot_000.pdf
  • Statistical Analysis Plan (2021-05-13): https://cdn.clinicaltrials.gov/large-docs/85/NCT03654885/SAP_001.pdf